## 伦理审查批件

## Approval Notice Template

项目编号: 2020BZYLL0902

项目名称:"慢痞消"治疗慢性萎缩性胃炎的临床研究

| 主要研究者:「霞 | 项目类别: 重点研发计划 |
|------------------|-------------------|
| 申办单位: 北京中医药大学科技处 | 合同研究组织 (CRO): |
| 审查类别: 初始审查 | 申查方式: 口快速申查 図会议审查 |
| 审查委员: 见附件 | 审查日期: 2020年12月28日 |

批准文件(注明版本号及日期),研究方案(版本号: V2.0,版本日期: 2021.01.06) 知情同意书(版本号: V2.0, 版本目期: 2020.01.06)

审查依据:根据 CFDA 《药物临床试验质量管理规范》(2003年)、《医疗器械临床试验质量管理规范》 (2016年)、世界医学会《赫尔辛基宣言》(2013年)、国际医学科学组织委员会《人体生物医学研究 国际伦理指南》(2016年)、国家卫生计生委《涉及人的生物医学研究伦理审查办法》(第11号,2016) 答。

审查决定: 同意

注:

- 1、本批件自签发日期有效期一年,起止时间 2021 年 1 月 26 日至 2022 年 1 月 26 日,研究者必须严格使 用经审查同意的知情同意书和研究方案。
- 2、研究开始前,请申请人完成临床试验注册。
- 3、凡涉及中国人类遗传资源、需要报批的研究项目,需告知在获得中国人类遗传资源管理办公室批准后 才能开始。
- 4、研究过程中若变更主要研究者,对临床研究方案、知情同意书、招募材料等的任何修改,请申请人提 交修正案审查申请。
- 5、发生严重不良事件,请申请人及时提交严重不良事件报告。
- 6、请按照伦理委员会规定的年度/定期跟踪审查频率,申请人在截止日期前1个月提交研究进展报告。
- 7、研究纳入了不符合纳入标准或符合排除标准的受试者,符合中止试验而未让受试者退出研究。给予错 误治疗或剂量,给予方案禁止的合并用药等没有遵从方案开展研究的情况;或可能对受试者的权益/健康 以及研究的科学性造成不良影响等违背 GCP 原则的情况,请申办者/监查员/研究者提交违背方案报告。
- 8、申请人暂停或提前终止临床研究,请及时提交暂停/终止研究报告。

9、完成临床研究,请申请人提交结题报告。

主任委员口副主任委员口签字:

时 间: 2021年1月26日

会议地点:线上会议

北京中医药大学医学伦理委员会

本项目持续审查频率 3 个月 6 个月 212 个月

联系人: 秦灵灵(010)53911431